CLINICAL TRIAL: NCT06291922
Title: Home-Based Exercise Program Using Mobile Technology After Left Ventricular Assist Device Implantation
Acronym: MOVE-LVAD II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 853181; R01HL166621 (NIH)
Record Dates: First submitted 2024-02-19; First posted 2024-03-04 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: Left ventricular assist device; Exercise; Ventricular assist device; HeartMate 3 (HM3)
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): The exercise intervention focuses on walking and strengthening exercises with a standardized protocol to guide exercise prescription and exercise progression based on data obtained from the activity tracking watch and smartphone app.
  Interventions: Behavioral: Exercise Intervention
- Usual Care (Other): The usual care group will be encouraged to increase daily walking activity as they tolerate, while complying with any activity restrictions from their clinical team. The Physical Activity Guidelines for Americans recommend increasing daily walking activity as tolerated to an average of 30 minutes daily, 5 times a week.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Exercise Intervention — See arm description.
  Arms: Exercise Intervention
Behavioral: Usual Care — See arm description.
  Arms: Usual Care

SUMMARY:
The goal of this clinical trial is to evaluate the effects of a home-based exercise program using mobile technology on physical activity and capacity, frailty and muscle mass, and quality of life in patients with a newly implanted HeartMate 3 left ventricular assist device (HM3 LVAD). Researchers will compare the effects of an exercise intervention vs. usual care on physical activity and capacity, frailty and muscle mass, and quality of life.

DETAILED DESCRIPTION:
Eligible subjects who sign the consent form will be randomized to either the exercise intervention arm or the usual care arm. As part of the baseline assessment, all subjects will measure their average daily steps during week 1 using a Garmin activity tracking watch, complete a six-minute walk test, complete frailty testing (including measurements of handgrip strength and gait speed), and complete surveys. Subjects will also complete a CT scan to evaluate muscle mass. After completing baseline assessments, subjects will be randomized to one of the study arms.

Subjects in the usual care arm will receive a Garmin activity tracking watch to wear continuously. Subjects will receive reminders from a smartphone app (Datos) to wear the watch. Subjects will be encouraged to increase daily walking as tolerated. In addition to standard of care clinic visits, they will receive phone calls from the study research coordinator reminding them to wear the watch and to walk.

Subjects in the exercise intervention arm will first have an initial training session with an interventionist to review exercises and safe practices. Subjects will receive an individualized exercise prescription for frequency, duration, and intensity of walking and strengthening exercises (including use of resistance bands and light weights). Subjects' progress in the exercise program will be remotely monitored using the activity tracking watch and the smartphone app, and subjects will complete questionnaires through the app. Subjects will complete video calls with the interventionist throughout the duration of the study and will receive updated personalized exercise prescriptions based on their progress.

Subjects in both study arms will have regular follow up VAD Clinic appointments per standard of care practices. Subjects will complete questionnaires, complete six-minute walk testing, complete frailty testing (including measurements of handgrip strength and gait speed), and undergo a chest CT scan without contrast as part of follow up activities. Throughout the study, data will be collected from the medical record.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Newly implanted with a HeartMate 3™ LVAD for the first time
3. Able to ambulate independently (with or without the use of an assistive device)
4. Owns a smartphone with Internet connection
5. Patient will be discharged home with LVAD or patient will be living at home with LVAD within 45 days of index discharge

Exclusion Criteria:

1. Major comorbidities or limitations that may interfere with exercise training (including significant orthopedic/neurologic limitations, decompensated heart failure, uncontrolled arrhythmias, unstable angina)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Effects of exercise intervention on physical activity and capacity (step count) | 6 months
  The investigators will compare the effects of the exercise intervention vs. usual care on physical activity and capacity measured by daily steps captured by an activity tracking watch.
Effects of exercise intervention on physical activity and capacity (distance) | 6 months
  The investigators will compare the effects of the exercise intervention vs. usual care on physical activity and capacity measured by six-minute walk test distance.

SECONDARY OUTCOMES:
Effects of exercise intervention on frailty and muscle mass (frailty status) | 6 months
  The investigators will compare the effects of the exercise intervention vs. usual care on frailty and muscle mass by evaluating frailty status (number of abnormal Fried frailty criteria, including handgrip strength).
Effects of exercise intervention on frailty and muscle mass (muscle quantity) | 6 months
  The investigators will compare the effects of the exercise intervention vs. usual care on frailty and muscle mass by evaluating muscle quantity (pectoralis muscle assessed by chest computed tomography scan).
Effects of exercise intervention on quality of life | 6 months
  The investigators will compare the effects of the exercise intervention vs. usual care on quality of life measured by the Kansas City Cardiomyopathy Questionnaire-12.
Cost-effectiveness of the exercise intervention vs. usual care | 6 months
  The investigators will determine the cost-effectiveness of the exercise intervention vs. usual care

CONTACTS AND LOCATIONS:
Overall Officials: Himabindu Vidula, MD, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - Henry Ford Health, Detroit, Michigan
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah Health, Salt Lake City, Utah